CLINICAL TRIAL: NCT05189002
Title: A Multicenter Randomized Double-blind Placebo-controlled Prospective Study to Evaluate the Safety and Efficacy of the Direct Factor Xa Inhibitor Dimolegin (DD217) in Prevention of Venous Thromboembolic Complications During Knee Replacement
Brief Title: A Study to Evaluate Dimolegin in Prevention of Thromboembolic Complications During Knee Replacement
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PharmaDiall Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AM217-02
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2021-12

CONDITIONS: Venous Thromboembolism
Keywords: Dimolegin; Dioxaban; DD217; factor Xa Inhibitor; anticoagulant; therapeutic anticoagulation; thromboprophylaxis; thrombosis; venous thromboembolism; knee replacement; anticoagulation
MeSH Terms: conditions — Venous Thromboembolism; Thrombosis | interventions — (+-)-(1'R*,2'S*,6'R*)-(2-hydroxy-4,6-dimethoxyphenyl)(3'-methyl-2'-(3''-methylbut-2''-enyl)-6-phenylcyclohex-3'-enyl)methanone; Dalteparin

STUDY DESIGN:
Intervention Model Description: Multicenter, double blind, randomized, prospective
Who Masked: Participant, Care Provider, Investigator
Masking Description: Dose Dimolegin - DD217 in each group was blinded for a patient and investigator (double-blind method) using six tablets for each administration, some of them contained Dimolegin - DD217, and others were masked as Placebo of the study product
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1a (Experimental): Patients from groups 1a took the study product once a day in doses 40 mg per os and saline solution subcutaneously. Dose was blinded for a patient and investigator (double-blind method) using six tablets for each administration, some of them contained Dimolegin - DD217, and others were masked as Placebo of the study product.
  Interventions: Drug: Dimolegin 40 mg
- Group 1b (Experimental): Patients from groups 1b took the study product once a day in doses 60 mg per os and saline solution subcutaneously. Dose was blinded for a patient and investigator (double-blind method) using six tablets for each administration, some of them contained Dimolegin - DD217, and others were masked as Placebo of the study product.
  Interventions: Drug: Dimolegin 60 mg
- Group 2 (Active Comparator): Patients from the control group (group 2) were received Fragmin in accordance with the instruction for medical use (5000 IU s/c once a day with 24-hour interval) and six Placebo tablets masked as study product Dimolegin - DD217 once a day.
  Interventions: Drug: Fragmin

INTERVENTIONS:
Drug: Dimolegin 40 mg — Dimolegin - DD217 - 40 mg
  Other Names: DD217
  Arms: Group 1a
Drug: Dimolegin 60 mg — Dimolegin - DD217 - 60 mg
  Other Names: DD217
  Arms: Group 1b
Drug: Fragmin — Fragmin 5000 IU in 0.2 ML Prefilled Syringe
  Other Names: Dalteparin sodium
  Arms: Group 2

SUMMARY:
This study is a multicenter, double-blind, randomized, prospective phase 2 dose ranging study to evaluate the safety and efficacy of Dimolegin - DD217 in prevention of venous thromboembolic complications in patients underwent knee replacement.

The study model is at each stage in parallel groups. Dimolegin - DD217 efficacy and safety in prevention of venous thromboembolic complications during knee replacement in groups of 80 patients will be investigated.

Patients who meet all inclusion criteria and none of the exclusion criteria will be randomized into three therapy groups: two therapy groups of the test drug Dimolegin - DD217 (40 mg (group 1a) and 60 mg (group 1b)) and one reference group (Fragmin).

Bilateral phlebography (preferably) or ultrasound duplex scanning (USDS) will be performed on the Day of the V13 visit.

It is planned to randomize 240 patients (160 patients in two different groups of Dimolegin - DD217 therapy and 80 patients in the reference group of Fragmin (INN: dalteparin).

The number of patients included in the study and randomized to receive Dimolegin - DD217, at the first stage, can be increased in the case of starting recruitment to additional group 1b.

The maximum number of patients who can be included in the study at the first stage is 320.

In total, no more than 480 patients can take part in the screening. Pharmacokinetic (PK) and pharmacodynamic (PD) parameters will be determined in patients who voluntarily give their consent to participate in the pharmacokinetic study (PKS) and pharmacodynamic study (PDS) and sign a Patient Information Leaflet with an informed consent form for participation in the PKS and PDS.

PK parameters are planned to be determined in 18-20 patients (50 % of each sex) in each patient group. Participation in the voluntary part of PK study will be offered to all patients.

The analysis of the composite endpoint frequency will be carried out using a generalized linear model for binary response.

A formal conclusion about superiority will be made if the lower limit of the specified confidence intervals exceeds the value of 0.0.

A formal conclusion on non-inferiority will be made if the lower limit of the specified confidence intervals exceeds the value of -0.05 (-5.0 %).

DETAILED DESCRIPTION:
This study is a multicenter, double-blind, randomized, prospective phase 2 dose ranging study to evaluate the safety and efficacy of Dimolegin - DD217 in prevention of venous thromboembolic complications in patients underwent knee replacement.

The study model is at each stage in parallel groups. Dimolegin - DD217 efficacy and safety in prevention of venous thromboembolic complications during knee replacement in groups of 80 patients will be investigated.

If the power of statistical tests (at α = 0.05) after the evaluation of intermediate data is at least 80 %, and the hypothesis of non-inferiority or superiority of Dimolegin - DD217 in comparison with Fragmin is proved, the study will be completed.

If the power of statistical tests (at α = 0.05) is less than 80 %, the recruitment of patients will continue. The required number of patients will be calculated taking into account the results obtained earlier, but no more than 120 patients per group.

Patients who meet all inclusion criteria and none of the exclusion criteria will be randomized into three therapy groups: two therapy groups of the test drug Dimolegin - DD217 (40 mg (group 1a) and 60 mg (group 1b)) and one reference group (Fragmin).

Patients from Dimolegin - DD217 groups 1a and 1b will receive the test drug once a day at doses of 40 mg (group 1a) orally or 60 mg orally (group 1b) and saline solution (Fragmin placebo) subcutaneously. Dimolegin - DD217 dose in each group will be blinded for the patient and the Investigator (double-blind method) using six tablets for each dose, of which some will contain Dimolegin - DD217, and the rest will be blinded as test drug placebo.

Patients from the reference group (group 2) will receive Fragmin in accordance with the instructions for medical use (5,000 IU s.c. 1 time per day with interval of 24 hours) and six placebo tablets blinded as the Dimolegin - DD217 test drug 1 time per day.

The first study drug dose will be taken in the morning the day after the surgery (visit V1). Then the study drug will be taken orally once a day (in the morning) for 12 days until day D13.

Bilateral phlebography (preferably) or USDS will be performed on the Day of the V13 visit.

As a result, Dimolegin - DD217 efficacy and safety in prevention of venous thromboembolic complications in total knee replacement (TKR) compared with standard therapy with Fragmin will be investigated. The study of PD/PK properties and the analysis of safety parameters will allow for choosing the optimal doses of the drug in terms of efficacy for phase 3 clinical trial.

During the study, following the safety analysis (if the frequency of cumulative major and clinically significant minor bleedings is more than 25 %) and treatment efficacy (if non-inferiority of the lowest dose is statistically significantly proved with 90 % confidence), IDMC recommendations, one of the Dimolegin - DD217 groups can be closed, and subjects may start to be enrolled to the 20-mg dose (group 1b). If randomization to one of the Dimolegin - DD217 groups is terminated prematurely, patients who have yet to be randomized can be randomized either to an open group or to a new group with an even lower dose (20 mg). In this case, randomization will be adapted to maintain a balance in sample size between all Dimolegin - DD217 groups and reference group. Based on the recommendations of IDMC, the sample size for a certain dose of Dimolegin - DD217 can be increased, while the sample size for other doses will be reduced so that the maximum planned number of patients is not exceeded.

Patients will be closely monitored for expected outcomes. The main outcomes on efficacy and safety will be centrally considered in IDMC. Investigators will have to inform IDMC in a timely manner about the expected occurrence of efficacy and safety outcomes (if possible, within 24 hours, fill out a package of documents for expert review and send it to IDMC) and report these outcomes in the electronic case report form in a timely manner (if possible within 24 hours). The Expert Committee will check the quality of the documents, including checking the data completeness.

The analysis of pharmacokinetics and pharmacodynamics will be carried out using validated analytical methods.

It is planned to randomize 240 patients (160 patients in two different groups of Dimolegin - DD217 therapy and 80 patients in the reference group of Fragmin (INN: dalteparin).

The number of patients included in the study and randomized to receive Dimolegin - DD217, at the first stage, can be increased in the case of starting recruitment to additional group 1b.

The maximum number of patients who can be included in the study at the first stage is 320.

In total, no more than 480 patients can take part in the screening. The study population will consist of adult patients aged 18 years and older who need an elective primary unilateral TKR (cement or cementless replacement).

The study will consist of a screening period, a clinical phase of the study and a "follow-up" period. Screening (visit V0) and hospitalization - must be performed no later than 14 days before surgery.

The clinical phase of the study will consist of a period of knee arthroplasty surgery and standard thromboprophylaxis, a period of randomization (V1) and administration of the test drug and reference drug (including in-patient follow-up, sampling for PK and PD analysis and monitoring of adverse events (AEs) in hospital, V1-V13) and a subsequent follow-up period 1 and 4 weeks (V14, V15) after the V13 visit.

The duration of the in-patient period is at least 14 (± 1) days, the period of out-patient follow-up is 4 weeks ± 3 days. Total study duration will not exceed 60 days.

PK and PD parameters will be determined in patients who voluntarily give their consent to participate in the PKS and PDS and sign a Patient Information Leaflet with an informed consent form for participation in the PKS and PDS.

PK parameters are planned to be determined in 18-20 patients (50 % of each sex) in each patient group. Participation in the voluntary part of PK study will be offered to all patients.

PK parameters will be calculated by the model-independent method.

For PKS and PDS, blood sampling will be carried out:

* At randomization visit in fasting condition before the standard therapy administration;
* In 1; 2; 4; 5; 6; 8; 12 hours after taking the first drug dose at the V1 visit;
* At visit days V2-V12 - 2 points each. The first point is 5-30 minutes before test drug/reference drug administration. The second is 4 hours ± 5 minutes after receiving the test drug/reference drug.
* At visit days (V13, V14, V15) - 1 point each. Total: 33 points. The total volume of blood for PK and PD studies to be collected from a patient during the study will not exceed 165 mL.

The Independent Data Monitoring Committee (IDMC) will regularly (at least after each planned interim analysis) receive up-to-date information on the outcomes of the study (in particular, on the frequency of combined outcome in terms of efficacy and frequency of major bleeding in different treatment groups) and adverse events (related to the study drug). IDMC will provide recommendations on the continuation or termination of patients' enrollment into the study groups, as well as on the need to start enrollment into an additional group (1b).

The analysis of the composite endpoint frequency will be carried out using a generalized linear model for binary response. The model will include a categorical predictor "therapy group". The comparison will be performed by calculating simple contrasts. The Fragmin group will be selected as the reference category.

A formal conclusion about superiority will be made if the lower limit of the specified confidence intervals exceeds the value of 0.0.

A formal conclusion on non-inferiority will be made if the lower limit of the specified confidence intervals exceeds the value of -0.05 (-5.0 %).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and older who need elective primary total knee replacement (cement or cementless arthroplasty)
* Signed informed consent
* Ability to comply with all protocol requirements
* Patients' consent to use adequate methods of contraception throughout the study

Exclusion Criteria:

* Surgery for an acute fracture 4 weeks before screening; septic inflammation of the joint, revision of the prosthesis or the absence of one leg
* Venous thrombosis of any localization or a confirmed PE episode at the present time or in the medical history
* Heparin-induced thrombocytopenia or other thrombocytopathies currently or in the history, hemorrhagic diathesis
* Obvious coagulopathy ongoing or in the history of the patient or a blood relative
* Congenital thrombophilia according to the medical history (deficiency of antithrombin III, protein C, protein S, Leiden mutation of coagulation factor V, increased level of coagulation factor VIII, mutation of prothrombin G20210A)
* Active bleeding (intracranial, intraocular, nasal, digestive or other localization) at present or within 6 months prior to screening, high risk of bleeding
* Collection of at least one volume unit of donated blood (> 500 mL) or blood transfusion during the previous 12 weeks
* Surgery on the brain or spinal cord, spine, ophthalmic or major surgery or injury in the last 90 days
* Gastrointestinal tract disorders that can disrupt the absorption of the study drug (Crohn's disease, ulcerative colitis, irritable bowel syndrome)
* Acute gastric or duodenal ulcer, erosive gastritis with increased risk of bleeding
* Significant cardiovascular diseases ongoing or within 6 months prior to screening, including: chronic heart failure of class III or IV (according to the classification of the New York Heart Association), myocardial infarction, unstable angina, surgery on the heart and coronary vessels (including percutaneous coronary intervention with or without coronary artery stenting), significant diseases of the heart valves, hemodynamically significant cardiac arrhythmias, transient ischemic attack, ischemic or hemorrhagic stroke, uncontrolled hypertension
* Active liver disease (viral hepatitis B or C, cirrhosis of the liver) and biliary tract disease, with the exception of non-alcoholic steatohepatitis with normal levels of hepatic transaminases (ALT and AST)
* Nephrotic syndrome, significant kidney diseases with the events of nephrotic syndrome (decreased filtration renal function with decreased estimated glomerular filtration rate (eGFR) < 60 according to the MDRD formula (MDRD)
* Malignant neoplasms during the last 5 years (with the exception of basal cell carcinoma for which radical treatment was carried out).
* Positive test for HIV, syphilis, hepatitis B or C markers (HBsAg and Anti-HCV)
* Significant drug or alcohol abuse according to the Investigator in the history or currently
* The development of trophic disorders of the lower extremities that do not respond to medical treatment
* Any condition, in which, according to the Investigator, surgical intervention or anticoagulants are contraindicated
* Body mass index (BMI) less than 18.5 or more than 40 kg/m2. Body weight above 130 kg
* Systolic BP > 180 mmHg and/or diastolic BP >110 mmHg, reported with two consecutive measurements for 15-30 minutes
* Hemoglobin < 105 g/L in women or < 115 g/L in men
* Abnormal laboratory parameters of the coagulation system (platelets, activated partial thromboplastin time (APTT), international normalized ratio (INR) and D-dimer), which, according to the Investigator and Medical Expert of the study, cause suspicion of blood clotting or problems in the hemostasis system in the patient
* eGFR < 60 mL/min/1.73 m2 (by MDRD formula)
* ALT or AST > 2 x upper limit of normal (ULN) or total bilirubin > 1.5 x ULN
* Hypersensitivity or contraindications to Dimolegin - DD217, dalteparin sodium, unfractionated heparin or warfarin; pig tissue preparations, radiopaque preparations (for multislice spiral computed tomography (MSCT) with intravenous enhancing)
* The need for constant use of parenteral or oral anticoagulants (for example, patients with artificial heart valves, patients with atrial fibrillation who are indicated for warfarin therapy)
* Systemic therapy with azole group drugs (ketoconazole, fluconazole, etc.), as well as other CYP3A4 inhibitors 7 days before and during screening.
* Previous and concomitant therapy: taking antiplatelet drugs, therapy with vitamin K antagonists, therapy with unfractionated heparin, low molecular weight heparin (LMWH), direct oral anticoagulants, the use of NSAIDs should be stopped at least 7 days before the start of the study therapy, systemic therapy with strong CYP3A4 and P-glycoprotein inhibitors, systemic therapy with strong inducers of CYP3A4 and P-glycoprotein
* Women who are pregnant or breastfeeding
* Women planning pregnancy during a clinical trial (including women who received a positive pregnancy test result during screening or before taking the study drug)
* Women of childbearing potential (including non-sterilized surgically and in the postmenopausal period less than 2 years) who do not want or cannot use adequate methods of contraception throughout the study. Adequate methods of contraception include the use of a condom or diaphragm (barrier method) with spermicide
* Participation in another clinical trial currently or within 30 days prior to screening, use of any investigational drug for 30 days or 5 half-lives (which is longer) prior to screening
* Affiliation to the investigational site: close relatives of the Investigator, dependent persons (for example, an employee or a person studying at the investigational site)
* Inability to read or write; unwillingness to understand and follow the study protocol procedures; non-compliance with the regimen of treatment or procedures which, according to Investigator, may affect the study results or patient's safety and prevent the patient from further participating in the study; any other concomitant medical or serious mental conditions, which make the patient ineligible for the clinical study, restrict validity of the consent or may affect the patient's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The total venosus thromboembolism (VTE) index | 14 Days
  The frequency of composite endpoint, which includes:
  * Asymptomatic deep vein thrombosis (DVT) detected by bilateral phlebography (preferably) or USDS at Visit V13 (Day D14±1);
  * Objectively confirmed by phlebography, USDS, computed tomography or other method symptomatic or asymptomatic DVT before Visit V13 (Day D14±1) inclusive;
  * Non-fatal PE before Visit V13 (Day D14±1) inclusive;
  * Fatal PE before Visit V13 (Day D14±1) inclusive;
  * Unexplained death, in which pulmonary embolism (PE) cannot be excluded before the Visit V13 (Day D14 ± 1) inclusive.

SECONDARY OUTCOMES:
The total venosus thromboembolism (VTE) index (W6) | 6 Weeks
  The frequency of composite endpoint, including:
  * Symptomatic VTE, non-fatal PE, fatal PE, unexplained death, in which PE cannot be excluded before the Visit V15 (W6 ±3 days) inclusive;
  * Objectively confirmed by phlebography, USDS, computed tomography or other method symptomatic or asymptomatic DVT before Visit V15 (W6±3 days) inclusive.

OTHER OUTCOMES:
The frequency of cumulative major and clinically significant minor bleeding on Visits V1- V13 | 14 Days
  The frequency of cumulative major and clinically significant minor bleeding on Visits V1- V13 (Days D2-D14±1) - primary safety endpoint.
The frequency of cumulative major and clinically significant minor bleeding before Visit V15 | 6 Weeks
  The frequency of cumulative major and clinically significant minor bleeding before Visit V15 (W6±3 days) - secondary safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry A Napalkov, Professor, Study Chair — Department of Faculty Therapy No. 1 of the Sechenov University
Locations (15):
- Russia (15):
  - GAUZ Bryansk City Hospital No. 1, Bryansk
  - Federal State Budgetary Institution National Medical Research Center of Traumatology and Orthopedics named after Academician G.A. Ilizarov the Ministry of Health of the Russian Federation, Kurgan
  - A budgetary medical institution Kursk Regional Clinical Hospital of the Health Committee of the Kursk Region, Kursk
  - GBUZ of the city of Moscow City Clinical Hospital No. 1 named after NI Pirogova of the Moscow City Health Department, Moscow
  - Federal State Budgetary Scientific Institution Russian Scientific Center for Surgery named after Academician B.V. Petrovsky, Moscow
  - GBUZ Moscow GKB im. S.P. Botkin of the Department of Health of the city of Moscow, Moscow
  - GBUZ of the Moscow region MONIKI them. M.F. Vladimirsky, Moscow
  - FBUZ Privolzhsky District Medical Center FMBA, Nizhny Novgorod
  - FSBEI HE Privolzhsky Research Medical University of the Ministry of Health of the Russian Federation, Nizhny Novgorod
  - GBUZ Penza Regional Clinical Hospital named after N.N. Burdenko, Penza
  - Federal State Budgetary Educational Institution of Higher Education Ryazan State Medical University named after Academician I.P. Pavlova of the Ministry of Health of the Russian Federation, Ryazan
  - St. Petersburg GBUZ City Hospital of the Holy Martyr Elizabeth, Saint Petersburg
  - FGBUZ Samara Regional Clinical Hospital named after V. D. Seredavin, Samara
  - GBUZ of the Republic of Mordovia Mordovian Republican Central Clinical Hospital, Saransk
  - FSBI Federal Center for Traumatology, Orthopedics and Endoprosthetics of the Ministry of Health of the Russian Federation, Smolensk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tovbin DG, Tarasov DN, Malakhov DV, Tserkovnikova NA, Aybush AV, Drozd NN. The Development of New Low-Molecular-Weight Factor Xa Inhibitors that are Potential Anticoagulants. Curr Drug Discov Technol. 2022;19(1):e010921191770. doi: 10.2174/1568009621666210224104940. PMID 33655836
- [Background] Tarasov DN, Tovbin DG, Malakhov DV, Aybush AV, Tserkovnikova NA, Savelyeva MI, Sychev DA, Drozd NN, Savchenko AY. The Development of New Factor Xa Inhibitors Based on Amide Synthesis. Curr Drug Discov Technol. 2018;15(4):335-350. doi: 10.2174/1570163815666180215114732. PMID 29468977